CLINICAL TRIAL: NCT06829329
Title: A Randomized, Multi-center Phase II Study to Evaluate the Efficacy and Safety of AHB-137 in Treatment-naive Participants With CHB
Brief Title: Study to Evaluate the Efficacy and Safety of AHB-137 in Treatment-naive Participants With Chronic Hepatitis B (CHB)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ausper Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB-10-8008
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2024-12

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — nas

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AHB-137 and placebo (Experimental)
  Interventions: Drug: AHB-137; Drug: Placebo
- AHB-137 and Nucleos(t)Ide Analogue (NAs) (Experimental)
  Interventions: Drug: AHB-137; Drug: NAs

INTERVENTIONS:
Drug: AHB-137 — AHB-137 will be administered .
Drug: NAs — NAs will be administered.
  Arms: AHB-137 and Nucleos(t)Ide Analogue (NAs)
Drug: Placebo — Placebo will be administered .
  Arms: AHB-137 and placebo

SUMMARY:
The study is to evaluate the efficacy and safety of AHB-137 in CHB participants. The total duration of the study, including screening phase, treatment phase and follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Participants voluntarily participate in the study, and sign the Informed Consent Form (ICF) prior to screening, able to complete the study according to the protocol;
* Male or female participants aged 18-65 years old (including the boundary value) at the time of signing the ICF;
* Male participants weighed higher than 50 kg and female participants weighted higher than 50 kg, Body Mass Index (BMI) between 18 to 32 kg/m^2(inclusive);
* Participants with positive HBsAg or HBV DNA greater than or equal to (≥) 6 months prior to screening and has not received antiviral treatment with interferon or NAs ;
* At screening, ALT<3×upper limit of normal (ULN);
* Use effective contraception as required;
* HBV DNA within the specified range at screening;
* HBsAg was within the specified range at screening.

Exclusion Criteria:

* Clinically significant abnormalities except chronic HBV infection;
* Any clinically significant liver diseases;
* Participants with severe infection requiring systemic anti-infection treatment 1 month before enrollment;
* Active hepatitis C, HIV antibody positive, treponema pallidum antibody positive;
* Hepatobiliary neoplasm malignant;
* The laboratory examination results are obviously abnormal;
* History of vasculitis or signs and symptoms of potential vasculitis;
* Anti-neutrophil cytoplasmic antibodies (ANCA) was positive at screening.
* History of extrahepatic disease that may be related to HBV immune status;
* Administration of immunosuppressants within 3 months prior to screening, except for short-term use (≤2 weeks) or topical/inhaled steroids. Administration of immunomodulators (thymosin) and cytotoxic drugs within 6 months prior to the first study intervention or have a history of vaccination within 1 month prior to screening or planned administration during the study;
* History of malignancy within the past 5 years or the discovery of suspected tumors during the screening period;
* Any suspicion of drug component allergy, or allergic constitution (various drug and food allergy, and judged by the investigator to be clinically significant) in participants;
* Participants who have significant trauma or major surgery within 3 months before screening, or plan to perform surgery during the study;
* Blood donation or blood loss more than 400 mL within 12 weeks before screening; Blood transfusion; Blood donation or blood loss not less than 200 mL within 1 month before screening;
* Those who are participating in another clinical trial, or have not undergone a protocol-specified washout period prior to this study;
* Participants who have received any oligonucleotide or small molecule interfering ribonucleic acid (siRNA) drugs;
* Any other circumstances or conditions for which the investigator considers that the participants are inappropriate to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-10-21 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving HBsAg lower than limit of detection (LOD) (0.05 IU/mL) and HBV DNA lower than lower limit of quantitation (LLOQ). | Up to 24 weeks

SECONDARY OUTCOMES:
Proportion of participants achieving functional cure during 24 weeks after discontinuation of all CHB therapy. | Up to 48 weeks
Number of Participants With HBsAg<LOD (0.05 IU/mL) and the percentage of participants with different levels of HBsAg reduction compared with baseline. | Up to 48 weeks
Number of participants with HBV DNA<LLOQ and the percentage of participants with different HBV DNA reduction. | Up to 48 weeks
Proportion of participants achieving HBsAg<LOD and HBV DNA<LLOQ, with or without HBsAb | Up to 48 weeks
Serum levels of HBsAg, HBV DNA, HBV RNA, HBcrAg, HBsAb | Up to 48weeks
Changes of the score of hepatitis B quality of life instrument (HBQOL) compared with baseline | Up to 48 weeks
  The HBQOL consists of 31 items covering 7 dimensions: psychological well-being, anticipation anxiety, vitality, stigma, transmissibility, vulnerability and virus response. Response options range from 1 to 5 with higher scores indicating more severe impact of Hepatitis B than lower scores.
Percentage of participants who reached HBeAg negative | Up to 48 weeks
  Only for participants with HBeAg positive at baseline
Percentage of participants achieving HBeAg seroconversion | Up to 48 weeks
  Only for participants with HBeAg positive at baseline
Proportion of participants with ALT normailzation in absence of rescue therapy. | Up to 48 weeks
  Only for participants with abnormal ALT at baseline
Time of ALT normalization in absence of rescue therapy | Up to 48 weeks
  Only for participants with abnormal ALT at baseline
Safety: number of participants with treatment-emergent adverse events (TEAEs), treatment-related adverse events(TRAEs), serious adverse events (SAE) and clinically significant examination results | Up to 48 weeks
  Examination including laboratory examination, electrocardiogram (ECG) examination
Immunogenicity: number and percentage of participants with detectable anti-drug antibodies (ADA) | Up to 48 weeks
The pharmacokinetic profile of AHB-137: Maximum concentration (Cmax) of AHB-137 in plasma | Up to 48 weeks
The pharmacokinetic profile of AHB-137: Area under the concentration-time curve (AUC) of AHB-137 | Up to 48 weeks
Plasma concentrations of AHB-137 | Up to 48 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Third People's Hospital of Zhenjiang, Zhenjiang, Jiangsu
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No